CLINICAL TRIAL: NCT01469559
Title: A Phase IIa Dose Escalation Pilot Study to Investigate the Safety and Tolerability of Intranasal Insulin in Subjects With Diabetic Polyneuropathy.
Brief Title: Safety Study of Intranasal Insulin in Type 1 Diabetes and Diabetic Peripheral Neuropathy
Acronym: IIDPN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, DR. LAWRENCE KORNGUT, Medical Doctor, Neurologist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UCALG-IIDPN
Record Dates: First submitted 2011-11-08; First posted 2011-11-10 (Estimated); Last update posted 2012-08-10 (Estimated); Status verified 2012-08

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Insulin; Diabetic neuropathy; Intranasal administration; Pilot project
MeSH Terms: conditions — Insulin Resistance; Diabetic Neuropathies | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Novolin Toronto insulin (Active Comparator)
  Interventions: Drug: Novolin Toronto insulin
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Novolin Toronto insulin — Subjects randomized to active drug are provided with 20 IU BID of Novolin Toronto at randomization (week 5). The dosing is prescribed to be taken 30 minutes after the morning meal (breakfast) and 30 minutes after the evening meal (supper). Subjects are asked to consume their meals and take their doses of study treatment within the same time frame each day. Dose escalations occur every 2 weeks with the insulin increasing to 40 IU BID at week 7, then 80 IU BID at week 9. The study completes at week 11. The total treatment period is 6 weeks. The insulin is diluted with an amount of normal saline to provide a total volume in the study treatment vial to equal 1.1 milliliters.
  Arms: Novolin Toronto insulin
Drug: Normal saline — Subjects randomized to placebo are provided with 1.1 milliliters of normal saline at randomization (week 5). The study completes at week 11. The total treatment period is 6 weeks. The dosing is prescribed to be taken 30 minutes after the morning meal (breakfast)and 30 minutes after the evening meal (supper). Subjects are asked to consume their meals and take their doses of study treatment within the same time frame each day. The amount of normal saline in the study treatment vial (1.1 milliliters) is identical in volume to the active insulin being used in the study .
  Arms: Normal saline

SUMMARY:
The aim of this study is to evaluate the safety and tolerability of intranasal insulin in people with type 1 diabetes and diabetic peripheral neuropathy and to determine whether intranasal insulin is effective in slowing the progression of diabetic neuropathy.

DETAILED DESCRIPTION:
Diabetic polyneuropathy (DPN) is a common complication of human type I and II diabetes mellitus, identified in up to 50% of diabetic subjects regardless of age or type of diabetes. As the global burden of diabetes heightens due to an epidemic of type II diabetes, the prevalence of DPN will concurrently rise. Clinical features of DPN include loss of sensation, propensity towards traumatic wound formation, neuropathic pain, motor weakness and falls.

At this time there is no specific therapy to arrest or reverse DPN. Previous work has demonstrated not only an absolute reduction in plasma insulin levels in Type I diabetes but also in type II diabetics. At the present, therapy for neuropathic pain associated with DPN is available, but only targets symptom relief and is only partially effective.

Intranasal insulin administration is a novel approach to the treatment of diabetic polyneuropathy (DPN) based on robust basic science research. Intranasal insulin is currently being studied in other conditions and has completed Phase II in subjects with cognitive impairment and mild Alzheimer's disease. Intranasal administration of insulin results in increased penetration into the cerebrospinal fluid and the peripheral nervous system while avoiding systemic absorption. Lack of systemic absorption results in maintenance of normal blood glucose levels in normal healthy subjects.

The objectives of the current study are as follows:

1. Primary: To determine the safety and tolerability of intranasal insulin delivery in subjects with type 1 diabetes and DPN.
2. Secondary: To determine whether intranasal insulin is efficacious in slowing the progression of DPN.

This study is designed as a double-blind, placebo-controlled, randomized, controlled-dose escalation phase 2 pilot clinical trial.

The duration of the study for each subject is 11 weeks with 6 weeks of blinded study treatment. The study treatment is either active study drug (Novolin Toronto insulin) or placebo (normal saline).

The phases of the study are as follows:

1. Screening phase (3 weeks): Potential subjects undergo screening procedures to determine eligibility. Procedures include informed consent, review of medical history, anthropometric measures, vital signs, physical examination (including a neurological assessment), and bloodwork.
2. Baseline phase (2 weeks): Eligibility of subjects is confirmed and subjects commence collection of protocol-specified blood glucoses on a daily basis. Nerve conduction tests and corneal confocal microscopy is completed prior to the start of the next phase.
3. Treatment phase (6 weeks): Subjects commence the study treatment at the lowest protocol-specified dose. If assigned to Novolin Toronto insulin, this is 20 international units (IU) twice daily (BID). Return visits to the clinic occur every two weeks for dose escalation. The dose increase is 40 IU BID, then 80 IU BID. Subjects assigned to normal saline receive a volume equivalent to the total volume given to the subjects taking insulin. Visits during the treatment phase also include safety bloodwork, serial blood glucose measurements every 15 minutes for a 2 hour period, review of any hypoglycemia, adverse events, changes to concomitant medications, assessment of neuropathy, questionnaires, teaching, and study treatment accountability/compliance assessment. The study completes at the 11 week time period, immediately prior to which the second nerve conduction study and corneal confocal microscopy is completed.

The study protocol is designed to monitor hypoglycemia throughout the baseline and treatment period for all subjects. Any severe hypoglycemia or significant increases in hypoglycemia (>30% compared to the baseline phase) will be reviewed by the Investigator on a case-by-case basis to determine continuation with study treatment. Any subject that undergoes discontinuation of study treatment will be continued to be followed to 11 weeks (without study treatment).

ELIGIBILITY:
Inclusion Criteria:

* Patients classified as having type 1 diabetes mellitus according to the Canadian Diabetes Association Criteria.
* Patients clinically defined as having DPN, meeting at least two of the following conditions:

  1. clinical signs of polyneuropathy;
  2. Symptoms of nerve dysfunction;
  3. Nerve conduction deficits in at least 2 nerves.
* Aged 18 through 70 years (inclusive).
* Body Mass Index (BMI) <30 kilograms/meter2.

Exclusion Criteria:

* Any other possible etiology contributing to the neuropathy:

  1. History of prolonged untreated hypothyroidism.
  2. Presence of untreated B12 deficiency.
  3. Presence of a paraproteinemia, detected using serum protein electrophoresis with a minimal threshold detection of 2 g/L.
  4. Use of a neurotoxic medication with a clear association with peripheral neuropathy within the past 1 year based upon clinical impression of association.
  5. Previous exposure chemotherapeutic agents with a clear association with peripheral neuropathy at any time.
* History of 2 or more severe hypoglycemic episodes within the previous 6 months.
* History of clustering of hypoglycemia episodes within the previous 12 months.
* History of active or recent (<5 years) malignancy.
* History of systemic or local nasal disease that would complicate the use of intranasal insulin.
* Presence of diabetic nephropathy requiring dialysis.
* Presence of active proliferative retinopathy requiring surgery within 6 months.
* Pregnancy or lactation (female subject of reproductive age must be on contraception).
* Active cardiovascular disease:

  1. Recent angina (<5 years)
  2. Recent myocardial infarction (<5 years)
  3. Congestive heart failure
* Active psychiatric disorder or previous history of psychosis.
* Unable to understand or provide consent.
* Previously documented hypersensitivity to insulin.
* History of hypoglycemia unawareness.
* Glycated hemoglobin < 7.0%.
* Ongoing involvement in another investigational drug trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-08; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Hypoglycemia monitoring | 8 weeks
  Hypoglycemia is defined by the development of autonomic or neuroglycopenic symptoms, and with or without the presence of a blood glucose measurement.
  All qualifying subjects are provided with blood glucose testing supplies to monitor blood glucoses six times daily from week 3 to week 11 of the study.
  Any severe hypoglycemia or increase of hypoglycemia of greater than 30% from the baseline phase (week 3 to week 5) is deemed clinically significant and is reviewed by the investigator to determine subject continuation with study treatment.

SECONDARY OUTCOMES:
Treatment satisfaction questionnaire for medication (TSQM) | 6 weeks
  The TQSM assesses the overall global impression of the treatment by the study subjects. During the study, the TSQM is administered at weeks 7, 9 and 11.
Adverse effects | 11 weeks
  The subject's overall health is assessed throughout the study to determine any changes with respect to existing history, in addition to capturing any new medical conditions that may arise.
The UTAH early neuropathy scale | 6 weeks
  The UTAH early neuropathy scale, a standarized physical examination scale, is used to measure changes in sensory neuropathy. During the study, the scale is administered at the time of randomization (week 5), then every 2 weeks until the end of study (week 11).
Corneal confocal microscopy | 6 weeks
  The corneal confocal microscopy measures corneal nerve fiber branch length and density. This procedure is done prior to week 5 (randomization) and immediately prior to week 11 (end of study).
Electrophysiology | 6 weeks
  The following components will be measured to monitor changes in nerve conduction:
  1. Sural conduction velocity
  2. Radial SNAP amplitude
  3. Radial:Sural SNAP ratio
  The nerve conduction tests are completed prior to week 5 (randomization) and immediately prior to week 11 (end of study).
McGill pain questionnaire | 6 weeks
  The McGill pain questionnaire, a standardized scale of rating pain on a scale of 0 (no pain) to 10 (worst pain), is used to monitor change in subject's pain symptoms. During the study, subjects complete this questionnaire at week 5 (randomization) and then every 2 weeks until the end of study (week 11).
Short Form-36 (SF-36) Quality of life scale | 6 weeks
  The SF-36 qualify of life scale, a standardized scale, is used to monitor change in subject reported functionality, well being, and overall health status. During the study, subjects complete this questionnaire at week 5 (randomization) and then every 2 weeks until the end of study (week 11).

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence M Korngut, MD, FRCPC, Principal Investigator — University of Calgary
Locations (1):
- Heritage Medical Research Clinic, Calgary, Alberta, Canada